CLINICAL TRIAL: NCT05915182
Title: A Real-world, Multicenter, 52-week Prospective Cohort Study to Capture the Reasons for Switch to Triple Combination Therapy and to Assess the Clinical and Patient Reported Outcomes in Adults With Moderate to Severe COPD Treated With Trixeo Aerosphere™ in Routine Care Settings in Greece.
Brief Title: Real-world, 52-week Prospective Study to Capture the Reasons for Switch to Triple Combination Therapy, Assess the Clinical and Patient Reported Outcomes in Adults With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Treated With Trixeo Aerosphere™ in Routine Care Settings in Greece
Acronym: TRIAENA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00082
Record Dates: First submitted 2023-05-28; First posted 2023-06-22 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD)
Keywords: Pulmonary Disease, Chronic Obstructive, Budesonide Glycopyrronium bromide Formoterol fumarate
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Combination Product: Budesonide Glycopyrronium bromide Formoterol fumarate pressurized Metered Dose Inhaler — Participants with moderate to severe Chronic Obstructive Pulmonary Disease

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a debilitating and progressive respiratory condition characterized by irreversible airflow limitation. The overall 5-year survival for COPD patients is 56-92%, depending on disease severity. Considering the recent introduction of the Budesonide, Glycopyrronium bromide and Formoterol fumarate Metered-Dose Inhaler (BGF MDI) in COPD therapeutic arsenal as well as the increasingly important role of real-world (RW) data in health care decisions, as it bridges gaps not addressed by randomized clinical trials, there is a need for RW evidence studies that can serve as inputs for Health Technology Assessment (HTA) submissions. In view of this need, this study is designed to generate RW evidence on the clinical and patient-reported outcomes of treatment with BGF MDI over a 52-week treatment period in routine care settings in Greece as well as to shed light on the reasons for switching from dual to triple therapy with BGF MDI, aiming at further characterizing the multifactorial aspects of inadequate COPD management that lead physicians to step-up treatment. The study is mainly descriptive in nature and is not planned to reject or affirm any formal statistical hypothesis. This is a single-country, non-interventional, multicenter, 52-week prospective cohort study, mainly based on primary data collection, which will include adult patients with moderate to severe COPD newly prescribed maintenance treatment with BGF MDI in routine care settings of Greece. This study design has been selected on the basis that such studies essentially, through collecting data generated in the course of routine clinical care about management practices and their outcomes from both the physician and patient perspective, help to bridge the knowledge gap between clinical research in controlled randomized settings and daily clinical practice. In line with the purely observational and non-interventional nature of the study, no changes to the current standard of care will be required and all aspects of treatment and clinical management of patients will be in accordance with local clinical practice and at the discretion of the participating physicians. The conduct of this study will adhere to the applicable national regulatory requirements governing the conduct of such type of clinical research. In addition, the study has been designed and will be conducted and reported in accordance with the ethical principles laid down in the Declaration of Helsinki, the Guidelines for Good Pharmacoepidemiology Practice (GPP) of the International Society for Pharmacoepidemiology, the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines where applicable, the European Union (EU) General Data Protection Regulation (GDPR), and the local rules and regulations. Patients will have been prescribed BGF MDI (Trixeo Aerosphere™) prior to informed consent (IC) obtainment and will be treated according to the local prescribing information (Summary of Product Characteristics [SmPC]) of the study medication and routine medical practice in terms of visit frequency and type of assessments performed. The assignment of the patient to this therapeutic strategy is not decided in advance by the study protocol but falls within current practice and the prescription of BGF MDI is clearly separated from the physician's decision to include the patient in the current study. In addition, every medical decision including the course of treatment will reflect exclusively the decision of the treating physician in a routine clinical situation according to the product's SmPC. Follow-up visit frequency will be determined by the treating physician, however study-related data will be collected at study enrollment and at 12, 24, 36, and 52-week data collection timepoints post-index (i.e., after BGF MDI treatment initiation) with an allowable time window of ±2 weeks for each data collection timepoint. Data collection at the aforementioned timepoints will be performed in the context of on-site routine visits at the private practices/hospital clinics. In addition, a telephone contact will take place at 4 (±1) weeks post-index for the sole purpose of administering COPD Assessment Test (CAT) by phone interview with the patient. Any visits/contacts occurring at other times not pre-planned in the context of the study will not be captured for the purposes of this study, except for safety-related information, exacerbation data, information on BGF MDI and concomitant COPD-related treatments, that will be collected on a continuous basis. Data collection at all indicated timepoints will be performed in the context of on-site routine visits at the private practices/hospital clinics. There are no dose regimens or diagnostic procedures pre-defined within this study plan. Participation in this observational, real-life study and its documentation procedure will not affect the routine treatment situation in any way.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 40 to 80 years (inclusive) at the time of BGF MDI initiation.
* COPD diagnosis for at least 12 months before BGF MDI initiation in accordance with the definition by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2022 Report, as assessed per physician's routine practice or as documented in the patient's chart.
* Patients who have been prescribed but not yet initiated treatment with Budesonide Glycopyrronium bromide Formoterol fumarate pressurized Metered Dose Inhaler (BGF MDI) according to the Summary of Product Characteristics (SmPC) and local market reimbursement criteria. Prescription of BGF MDI must have occurred prior to signed Informed Consent (IC) and the decision to prescribe this therapy must by clearly separated from the physician's decision to include the patient in the current study.
* Spirometry-determined moderate to severe disease defined as post-bronchodilator (post-BD) Forced Expiratory Volume in 1 Second (FEV1)/Forced vital capacity (FVC) ratio <0.70 and FEV1 <80% predicted normal value based on most recent spirometry performed within the 3-month period prior to BGF MDI initiation.
* Current or former conventional cigarette smokers with a history of at least 10 pack-years of smoking.
* Patients must be able and willing to read and to comprehend written instructions, and to comprehend and complete the questionnaires required by the protocol.
* Patients must provide a written IC prior to inclusion to the study.

Exclusion Criteria:

* COPD due to documented α-1 antitrypsin deficiency.
* Subjects with current diagnosis of active tuberculosis, lung cancer or lung metastasis, significant bronchiectasis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension, interstitial lung diseases or other active clinically significant pulmonary diseases.
* Subjects with other uncontrolled disease.
* Recent (≤3 months) major cardiac or pulmonary event (for example myocardial infarction, pulmonary embolism).
* Respiratory tract infection [including, among others, Coronavirus Disease 2019 (COVID-19)] that has not resolved ≤30 days prior to BGF MDI initiation.
* Requirement of long term (at least 15 hours daily) oxygen therapy.
* Current or recent (≤4 weeks prior to BGF MDI initiation) long-term chronic maintenance use of systemic corticosteroids or antibiotic treatment for any reason other than COPD.
* Current or recent (≤4 weeks prior to BGF MDI initiation) participation in the acute phase of a Pulmonary Rehabilitation Program.
* Currently pregnant (or intention to become pregnant), breastfeeding or lactating women.
* Participation in a non-interventional observational trial that might, in the investigator's opinion, influence the assessment for the current study, or participation in any interventional observational or clinical trial in the last 30 days prior to enrollment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population from private practices and hospital clinics specializing in the management of Chronic Obstructive Pulmonary Disease (COPD) in geographically diverse locations throughout Greece, with a balanced representation of public, academic and private sector in Greece
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the CAT total and item scores at 12 weeks post index | At 12 weeks after treatment initiation
  Assess the change in Chronic Obstructive Pulmonary Disease (COPD) health status measured by the COPD Assessment Test (CAT) in COPD patients initiated on Budesonide, Glycopyrronium bromide, Formoterol fumarate Metered Dose (BGF MDI) Inhaler after 12 weeks of treatment
Percentage of patients achieving a ≥ 2-point reduction from baseline in CAT total score at 12 weeks post index | At 12 weeks after treatment initiation
  Estimate the proportion of CAT responders among COPD patients initiated on Budesonide, Glycopyrronium bromide, Formoterol fumarate Metered Dose (BGF MDI) Inhaler after 12 weeks of treatment

SECONDARY OUTCOMES:
Frequency of reasons of switch from dual to triple combination therapy with BGF MDI in the overall study population | At treatment initiation timepoint
  To describe and count in numbers the reasons for switch from dual LAMA/LABA or ICS/LABA to single-inhaler triple combination therapy with BGF MDI
Change from baseline in the COPD Assessment Test (CAT) total and item scores at 4, 24, 36 and 52 weeks post index | At 4, 24, 36, 52 weeks after treatment initiation
  To assess the change in COPD health status measured by the CAT among COPD patients initiated on BGF MDI after 4, 24, 36, and 52 weeks of treatment
Percentage of patients achieving a ≥ 2-point reduction from baseline in CAT total score at 4, 24, 36, and 52 weeks post index | At 4, 24, 36, 52 weeks after treatment initiation
  To estimate the proportion of CAT responders among COPD patients initiated on BGF MDI after 4, 24, 36, and 52 weeks of treatment
Change from baseline in the St. George's Respiratory Questionnaire for COPD (SGRQ-C) total and component scores at 12 and 52 weeks post index | At 12, 52 weeks after treatment initiation
  To assess the change in HRQoL measured by the SGRQ-C on the overall study population, after 12 and 52 weeks of treatment
Percentage of patients achieving a ≥ 4-point reduction from baseline in SGRQ-C total score at 12 and 52 weeks post index | At 12, 52 weeks after treatment initiation
  To assess the change in HRQoL measured by the SGRQ-C to estimate the proportion of SGRQ-C responders among COPD patients initiated on BGF MDI after 12 and 52 weeks of treatment.
Baseline Dyspnea Index (BDI) focal and domain scores at baseline | At treatment initiation timepoint
  To assess the severity of dyspnea at baseline measured by the baseline dyspnea index (BDI)
Transition Dyspnea Index (TDI) focal and domain scores at 12, 52 weeks post index | At 12, 52 weeks after treatment initiation
  To estimate the change in dyspnea severity (measured by the TDI) on the overall study population after 12 and 52 weeks of treatment.
Percentage of patients achieving a TDI focal score ≥ 1 unit at 12 and 52 weeks post index | At 12, 52 weeks after treatment initiation
  To estimate the proportion of TDI responders among COPD patients initiated on BGF MDI after 12 and 52 weeks of treatment
Change from baseline in pre dose trough Forced Expiratory Volume in 1 Second (FEV1) at 12, 24, 36, and 52 weeks post index | At 12, 24, 36, 52 weeks after treatment initiation
  To assess the change in spirometric lung function as measured by FEV1 on the overall study population after 12, 24, 36, and 52 weeks of treatment
Percentage of patients with increase from baseline in pre dose trough FEV1 ≥100 mL at 12, 24, 36, and 52 weeks post index | At 12, 24, 36, 52 weeks after treatment initiation
  To estimate the proportion of FEV1 responders among COPD patients initiated on BGF MDI after 12, 24, 36, and 52 weeks of treatment
Percentage of patients achieving the Minimum Clinically Important Difference (MCID) in pre dose trough FEV1 and in at least one Patient Reported Outcome (PRO) (SGRQ, CAT, or TDI) at 12 weeks post index | At 12 weeks after treatment initiation
  To determine the Early Clinically Important Improvement (ECII) rate in COPD patients initiated on BGF MDI after 12 weeks of treatment
Percentage of patients achieving the MCID in pre dose trough FEV1 and in at least one PRO (SGRQ, CAT, or TDI) at 52 weeks post index among the 12 week Early Clinically Important Improvement (ECII) responders | At 52 weeks after treatment initiation
  To assess the CII rate after 52 weeks of treatment among the 12-week ECII responders
Number of moderate and severe exacerbations that occurred during the 52 week period before the index date | At treatment initiation timepoint
  To describe the number of moderate and severe exacerbations during the 52 week period prior to BGF MDI initiation
Number of moderate and severe exacerbations that occurred during the 52 week period after the index date | During 52 weeks after treatment initiation
  To describe the number of moderate and severe exacerbations during the 52-week period after BGF MDI initiation
Percentage of patients achieving (a) the MCID in pre dose trough FEV1, (b) the MCID in at least one PRO, (c) at least 50% reduction in COPD moderate/severe exacerbations or exacerbation free state at 52 weeks post index | At 52 weeks after treatment initiation
  To assess the overall treatment response rate based on lung function, PROs and exacerbation rate after 52 weeks of treatment with BGF MDI
Percentages of patients achieving each of the aforementioned individual response measures as well as their combinations at 52 weeks post index | At 52 weeks after treatment initiation
  To assess the response rates based on individual measures of lung function, PROs, and exacerbation rate after 52 weeks of treatment with BGF MDI
Treatment Satisfaction Questionnaire for Medication version II (TSQM vII) scores at 12 weeks post index | At 12 weeks after treatment initiation
  To evaluate the treatment satisfaction, assessed by the Treatment Satisfaction Questionnaire for Medication (TSQM vII) after 12 of treatment with BGF MDI
TSQM vII scores at 52 weeks post index or at premature withdrawal from the study | At 52 weeks after treatment initiation
  To evaluate the treatment satisfaction, assessed by the Treatment Satisfaction Questionnaire for Medication (TSQM vII) after 52 weeks of treatment with BGF MDI
Single item score of Patient Global Impression of Change (PGIC) questionnaire at 52 weeks post index or at premature withdrawal from the study | At 52 weeks after treatment initiation
  To assess the patient-reported overall change in health status since the start of treatment with BGF MDI, using the Patient Global Impression of Change (PGIC) questionnaire
Single item score of Patient Global Impression of Severity (PGIS) questionnaire at 12, 24, 36 and 52 weeks post index | At 12, 24, 36, 52 weeks after treatment initiation
  To assess the patient-reported overall global impression of severity after 12, 24, 36, and 52 weeks of treatment with BGF MDI, using the Patient Global Impression of Severity (PGIS) questionnaire
Medication Adherence Report Scale (MARS-5) total score at 12, 24, 36 and 52 weeks post index | At 12, 24, 36, 52 weeks after treatment initiation
  To assess patients' adherence to treatment with BGF MDI, using the Medication Adherence Report Scale (MARS-5), after 12, 24, 36, and 52 weeks of treatment
Percentage of completely adherent (for example MARS-5 score=25) and not completely adherent patients (for example MARS-5 score: ≤ 24 points) at 12, 24, 36 and 52 weeks post index | At 12, 24, 36, 52 weeks after treatment initiation
  To assess the number of patients completely and not completely adherent at 12, 24, 36 and 52 weeks post-index
Percentage of patients remaining on treatment with BGF MDI at 52 weeks post index | At 52 weeks after treatment initiation
  To assess number of patients remaining on treatment at 52-weeks of treatment
Percentage of patients having discontinued treatment with BGF MDI at 52 weeks post index and description of reasons for treatment discontinuation | At 52 weeks after treatment initiation
  To assess the number of patients having discontinued treatment at 52 weeks of treatment
Time from the start of BGF MDI to all cause treatment discontinuation | During 52 weeks after treatment initiation
  To assess the time from the start of BGF MDI to all cause treatment discontinuation

CONTACTS AND LOCATIONS:
Locations (8):
- Greece (8):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Corfu
  - Research Site, Crete
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki